CLINICAL TRIAL: NCT00336973
Title: A Phase IV Open-Label Study to Evaluate the Efficacy and Safety of 1.0 mg/kg Raptiva (Efalizumab) in Adult Subjects With Chronic Moderate or Worse Plaque Psoriasis Who Have Had an Inadequate Response to an Anti-TNF Agent
Brief Title: A Study to Evaluate Raptiva in Subjects With Chronic Moderate or Worse Plaque Psoriasis Who Have Had an Inadequate Response to an Anti-TNF Agent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACD3780g
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2009-06-05 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2009-04

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Raptiva; Anti-TNF
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: efalizumab

INTERVENTIONS:
Drug: efalizumab — Subcutaneous repeating dose

SUMMARY:
This is a Phase IV open-label study to evaluate the efficacy and safety of SC efalizumab in adult subjects (18 years of age and older) with chronic moderate or worse plaque psoriasis who have had an inadequate response to treatment with an anti-TNF agent. The study will consist of a screening period, a treatment period, and an observation period. All subjects will begin in the screening period (the length of which is dependent on the previous anti-TNF agent treatment). Approximately 100 eligible subjects will receive treatment from Day 0 through Day 168.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic (6 months or greater) moderate or worse plaque psoriasis
* Have had an inadequate response to at least 12 weeks of treatment with an anti-TNF agent, where an inadequate response is defined as: PGA ratings of moderate (3), severe (4), or very severe (5), and BSA involvement of 5% or greater
* Be a candidate for systemic therapy or phototherapy in the opinion of the investigator
* Be naive to efalizumab treatment
* Weigh no more than 200 kg
* For women of childbearing potential, use a method of contraception acceptable to the investigator to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study and for 6 weeks after the last dose of efalizumab

Exclusion Criteria:

* Have a history of psoriatic arthritis that meets one of the following criteria: Is not controlled with non-steroidal anti-inflammatory drugs (NSAIDs);Requires the use of disease modifying antirheumatic drugs (DMARDs), including biologics while enrolled in the study; Please note that if, following enrollment, a subject requires treatment with a DMARD, study drug treatment should be discontinued and the subject should be moved into the observation period of the study. The subject should have the observation period assessments performed at the appropriate intervals as per the protocol
* Have a history of hypersensitivity to efalizumab or any of its components
* Are using any excluded therapy
* Are currently abusing alcohol or illegal drugs
* Have a history of or an ongoing uncontrolled serious bacterial, viral, fungal, or atypical mycobacterial infection. This includes diagnoses that required more than 2 weeks of therapy, such as endocarditis and osteomyelitis, which have been treated in the past 6 months. In addition, if the subject is currently receiving antibiotics, antivirals, or antifungals for an infection or for suppression or prophylaxis for any diagnosis, the subject will be excluded.
* Have any history of opportunistic infections (e.g., systemic fungal infections, parasites)
* Are seropositive for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus (HIV). Subjects will undergo testing during screening, and any subjects who are seropositive for hepatitis B antigen, hepatitis C antibody, or HIV will be excluded.
* Have a history of active tuberculosis or are currently undergoing treatment for tuberculosis. A purified protein derivative (PPD) test will be performed at the screening visit. Subjects with a positive PPD test (not due to BCG vaccination) or chest x-ray will be excluded.
* Have the presence or history of malignancy, including lymphoproliferative disorders. Subjects with a history of fully resolved basal or squamous cell skin cancer may be enrolled.
* Are pregnant or lactating women
* Have a diagnosis of hepatic cirrhosis, regardless of cause or severity
* Have a history of thrombocytopenia
* Have a history of clinically significant hemolytic or unexplained anemia
* Have been exposed to any experimental drugs or treatments within 30 days or 5 half-lives, whichever is longer, prior to the screening visit
* Have had any previous exposure to efalizumab
* Have been vaccinated with a live virus or live bacteria within the 14 days prior to the first dose of efalizumab
* Have any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug or would significantly interfere with the subject's ability to comply with the provisions of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Efalizumab: After an initial conditioning dose of 0.7 mg/kg of subcutaneous (SC) study drug on Day 0, participants received 23 weekly doses of 1.0 mg/kg of SC study drug beginning on Day 7
Period: Overall Study
Arm/Group | Efalizumab
Started | 66
Completed | 33
Not Completed | 33

BASELINE CHARACTERISTICS:
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Physician's Global Assessment (PGA) Rating of Clear (0), Almost Clear (1), or Mild (2)
Description: The PGA scale used in this study was: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe
Time Frame: Day 84
Population: Intent-to-treat (ITT)
Measure: Number; unit: percentage
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
percentage | 34.8 [0.235 to 0.476]

2. Secondary Outcome: Proportion of Subjects With a PGA Rating of Clear (0), Almost Clear (1), or Mild (2)
Description: The PGA scale used in this study was: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe
Time Frame: Day 168
Population: Intent-to-treat (ITT)
Measure: Number; unit: percentage
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
percentage | 31.8 [0.209 to 0.444]

3. Secondary Outcome: Proportion of Subjects With a PGA Rating of Clear (0) or Almost Clear (1)
Description: The PGA scale used in this study was: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe
Time Frame: Day 84
Population: Intent-to-treat (ITT)
Measure: Number; unit: percentage
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
percentage | 9.1 [0.034 to 0.187]

4. Secondary Outcome: Proportion of Subjects With a PGA Rating of Clear (0) or Almost Clear (1)
Description: The PGA scale used in this study was: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe
Time Frame: Day 168
Population: Intent-to-treat (ITT)
Measure: Number; unit: percentage
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
percentage | 21.2 [0.121 to 0.330]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other